CLINICAL TRIAL: NCT03195504
Title: Effectiveness of Apneic Oxygenation Using High-flow Nasal Cannula in Morbidly Obese Patients Undergoing General Anesthesia
Brief Title: High-flow Nasal Oxygenation in Obese Patients During Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, David Wong, Professor Anesthesia (MD), University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-6264.0
Record Dates: First submitted 2017-06-05; First posted 2017-06-22 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Apneic Oxygenation; High-flow Nasal Cannulae; Bariatric Surgery; Anesthesia Induction

STUDY DESIGN:
Intervention Model Description: Consented patients will be randomly assigned either to the interventional group (High Flow Nasal Cannula- HFNC) or to the control group (CON). The Group HFNC will be preoxygenated using HFNC and the Group CON will receive standard preoxygenation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC (High Flow Nasal Cannulae) (Experimental): High Flow Nasal Cannulae providing humidified, high-flow oxygen during induction of anesthesia
  Interventions: Device: HFNC
- CON (control) (Active Comparator): Standard flow oxygen during induction of anesthesia
  Interventions: Device: CON (control)

INTERVENTIONS:
Device: HFNC — High flow nasal oxygen (60 l) under GA
  Arms: HFNC (High Flow Nasal Cannulae)
Device: CON (control) — Standard oxygen (10-15 l) under GA
  Arms: CON (control)

SUMMARY:
Before going off to sleep patients are given oxygen to saturate blood with oxygen to extend time before a decrease in the level of oxygen in the blood occurs. During this period, obese patients have a faster decrease in the level of oxygen in their blood. This study uses a device called "high-flow nasal cannula" (HFNC), which delivers humidified high-flow oxygen through 2 small plastic tubes placed just inside nostrils. In the intensive care unit settings this device has been used extensively and has become a standard practice. Purpose of this study is to determine whether these high-flow nasal cannula increase the time safely when going to sleep during elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age more than18 years old
* ASA status I-III
* Elective surgery performed under general anesthesia requiring endotracheal intubation
* BMI more than 40 kg/m2

Exclusion Criteria:

* Chronic respiratory disease
* SpO2 <98% after supplementing oxygen
* Previous or anticipated difficult intubation
* Uncontrolled hypertension
* Ischemic heart disease
* Congestive heart failure
* Increased intracranial pressure
* Uncontrolled GERD
* Known allergy or contraindication to anesthesia drugs
* Nasal blockade contraindicating the use of HFNC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Measurement of safe apnea time | Maximum up to 6 minutes
  Safe apnea time, defined by time to desaturation (SpO2 > 95%) or apnea maximum up to 6 minutes

SECONDARY OUTCOMES:
Highest EtCO2 | Every minute up to 5 minutes on commencing ventilation
  Highest EtCO2 on commencing ventilation
Lowest SpO2 | Every minute up to 5 minutes after intubation
  Lowest SpO2 during intubation procedure
Time to regain baseline SpO2 | Up to 5 minutes after intubation
  Time to regain baseline SpO2 after intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wong DT, Dallaire A, Singh KP, Madhusudan P, Jackson T, Singh M, Wong J, Chung F. High-Flow Nasal Oxygen Improves Safe Apnea Time in Morbidly Obese Patients Undergoing General Anesthesia: A Randomized Controlled Trial. Anesth Analg. 2019 Oct;129(4):1130-1136. doi: 10.1213/ANE.0000000000003966. PMID 31584919